CLINICAL TRIAL: NCT00174811
Title: Multinational, Randomized, Double-Blind, Double-Dummy, Comparative Study to Evaluate the Efficacy and Safety of Telithromycin 25 mg/kg Given Once Daily for 5 or 10 Days Depending on Age and Previous Treatment History Versus Cefuroxime Axetil 15 mg/kg, Given Twice Daily for 10 Days, in Children With Acute Otitis Media
Brief Title: Comparative Study to Evaluate the Efficacy and Safety of Telithromycin Given Once Daily Versus Cefuroxime Axetil Given Twice Daily in Children With Middle Ear Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pediatric development program terminated by sponsor
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6131; HMR3647B/3001
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Otitis Media
Keywords: acute otitis media; controlled clinical trial; telithromycin; cefuroxime axetil; middle ear infections; tympanocentecis
MeSH Terms: conditions — Otitis Media | interventions — telithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: telithromycin (HMR3647)

SUMMARY:
The clinical activity of telithromycin vs. cefuroxime in children with acute infections of the middle ear, ages 6 months to 59 months old will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥6 months and <59 months of age with AOM;
* Recent (within the last 72 hours) and rapid onset of AOM signs and symptoms;
* The presence of MEF on otoscopy indicated by a bulging tympanic membrane;
* Otalgia or ear tugging or touching within the last 24 hours that interferes with or precludes normal activity or sleep;
* At least 1 of the following clinical findings not specific to AOM: fever, vomiting, diarrhea, anorexia, sleep disturbance, or irritability;
* Tympanocentesis performed per protocol with MEF sample collected;
* Informed consent must be obtained in writing at enrollment into the study, from the child's parent/legally authorized representative. The parent/legally authorized representative has agreed to provide follow-up information and arrange for all scheduled visits, even in the event that study medication is discontinued.

Exclusion Criteria:

* Uncertain diagnosis of AOM or signs and symptoms of AOM that would make the subject a candidate for observation and analgesic therapy with observation for 2-3 days;
* Otorrhea or tympanostomy tube present in either ear at study entry;
* Otitis externa;
* Down syndrome, cleft palate, craniofacial disorders, cystic fibrosis/mucoviscidosis, immotile cilia syndrome, congenital immunodeficiency or acquired immunodeficiency syndrome with <25% CD4 count or requiring prophylaxis for Pneumocystis jiroveci (carinii) or requiring treatment for an opportunistic infection;
* Known congenital prolonged QT syndrome;
* Uncorrected hypokalemia (≤3 mmol/L [mEq/L]), hypomagnesemia (based on laboratory assessment), bradycardia (<50 bpm);
* Myasthenia gravis;
* Known impaired renal function, as shown by the creatinine clearance ≤25 mL/min;
* Any medical condition (including developmental disorders, visual disorders, or ocular abnormalities) that, in the opinion of the investigator, would interfere with implementation of the protocol or interpretation of the study results;
* The subject:
* Is being treated with drugs not permitted by the study protocol ie, cisapride, pimozide, astemizole, terfenadine, ergotamine, dihydroergotamine, class IA (eg, quinidine and procainamide) or Class III (eg, dofetilide) antiarrhythmic agents, simvastatin, lovastatin and atorvastatin;
* Is currently being treated with systemic antibacterials or has been treated with systemic antibacterials within 5 days prior to enrollment;
* Has been treated with any investigational medication within the last 30 days; or
* Has been treated with rifampicin, phenytoin, carbamazepine, or St. John's wort within the last 2 weeks.
* History of hypersensitivity or intolerance to macrolides, penicillins, or cephalosporins;
* Previous enrollment in this study or previous treatment with telithromycin;
* Children of the investigator or subinvestigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the protocol.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 639 (Actual)
Dates: Start 2005-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Clinical cure at the posttherapy/test-of-cure (TOC) Visit 3 (Day 13-17).

SECONDARY OUTCOMES:
Time to symptom resolution (TSR).
Clinical cure by protocol-defined causative pathogen isolated at baseline·
Bacteriological eradication in population with protocol-defined causative pathogen isolated at baseline.
Safety of telithromycin versus cefuroxime axetil.
Plasma telithromycin concentrations during treatment in the subpopulation of subjects participating in the pharmacokinetic (PK) substudy.
Health resource utilization and impact on usual activities.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi- Aventis Administrative Office, Paris, France